CLINICAL TRIAL: NCT01250626
Title: Establish the Caring Model of Children With Chronic Kidney Disease and End-stage Renal Disease: To Set up Childhood Glomerular Filtration Rate (GFR) Formula in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Ching-Yuang Lin, M.D.,PhD., China Medical University
Other Study IDs: DMR99-IRB-139
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-08

CONDITIONS: Chronic Kidney Disease; End-Stage Renal Disease
Keywords: Inulin; childhood GFR formula
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- a single-group study: Pediatric OPD, age < 18 y/o.

SUMMARY:
Inulin's usefulness as a diagnostic agent is based on the method of its elimination from the body. Inulin is biologically inert, unbound by plasma proteins, freely filtered at the glomerulus, and is neither reabsorbed, metabolized nor secreted by the kidneys. It is excreted almost entirely by glomerular filtration. Inulin clearance is considered to be identical to glomerular filtration rate (GFR).

ELIGIBILITY:
1. Main inclusion criteria: Pediatric OPD, age < 18 y/o.
2. Main exclusion criteria: Acute renal failure, edema, muscular dystrophy, pleural effusion, ascites, malnutrition, neurogenic bladder, heart failure and ketoacidosis. And taken cimetidine or trimethoprim, and accepted renal replacement therapy.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric OPD, age < 18 y/o.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-08